CLINICAL TRIAL: NCT05298410
Title: An Open Label Study to Investigate the Safety and Efficacy of an NAD+ Boosting Investigational Product Together With a Low Carbohydrate Diet in an Adult Population With Mild Hypertension and Eligible for Normal-standard-of-care
Brief Title: The Safety and Efficacy of an NAD+ Boosting Product Together With a Low Carbohydrate Diet in Adults With Mild Hypertension and Eligible for Normal-standard-of-care
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Limitless Research Inc. (Other)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19LPHL
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Hypertension
Keywords: NAD+ boosting investigational product; Mild hypertension; Limitless; Low carbohydrate diet
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Limitless (Experimental): Participants will be instructed to take Limitless capsules for 30 days starting with the first dose to be administered in clinic on Visit 2 (Day 1, Baseline). The last dose will occur in clinic on Visit 3 (Day 30). Participants will be instructed to take two capsules two hours with water after breakfast, and two capsules two hours after dinner. Do not take food after evening dose before bed. (i.e. no snacking or desserts.). If a dose is missed participants are instructed to skip that dose. Participants will be advised not to exceed four capsules daily.
  Interventions: Other: Limitless

INTERVENTIONS:
Other: Limitless — Participants will be instructed to take Limitless for 30 days.

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of Limitless, in combination with a low-carbohydrate diet, after 30 days of supplementation in an adult population. Changes from baseline to Day 30 post-supplementation on several parameters of vascular function will be examined and safety outcomes will be determined.

DETAILED DESCRIPTION:
With an aging population, and the resulting economic and health burdens, strategies to support healthy aging and mitigate age-associated metabolic changes are essential.

Recent studies have demonstrated that decreases in nicotinamide adenine dinucleotide (NAD+) levels in multiple tissues is involved in the pathogenesis of age-associated diseases. Therefore, strategies to support NAD+ levels and prevent the decline of NAD+ with age have drawn significant attention. NAD+ precursors have also been proposed to augment NAD+ and support healthy aging. While NAD+ precursors share some similarities, there are differences in their bioavailability and safety profiles. Both nicotinamide mononucleotide (NMN) and nicotinamide riboside (NR) are orally bioavailable and appear to increase NAD+ levels more efficiently than nicotinic acid (NA). Further, a study in rodents suggests that NMN is retained in the body longer than NA. Unlike NMN, NA is associated with several adverse effects such as cutaneous flushing and nausea and hepatoxicity in sustained release-formulations. Recently, the first clinical study examining the safety and bioavailability of NMN supplementation found that single orally administered doses of 100-500 mg were safe and well-tolerated.

The investigational product in this study contains NMN, in addition to berberine, R-lipoic acid, garlic powder, agmatine, black pepper extract, fisetin and L-citrulline malate. Preclinical studies have shown that restoring NAD+ levels by supplementation of NMN can ameliorate some of the functional defects caused by its decline. Further, there are numerous proof-of-concept in vitro and in vivo animal studies indicating that NMN supplementation has beneficial biological effects. Administration of 100 mg/kg/day of NMN for 12-months mitigated age-associated physiological declines in energy metabolism, insulin sensitivity, and plasma lipid profile while age-associated body weight gain was decreased. Other animal studies have shown that NMN supplementation improved glucose intolerance and lipid profiles in models of high-fat-induced and age-induced diabetic mice. Further, 300 mg/kg/day of NMN supplementation for 8 weeks in old mice ameliorated age-associated nitric oxide (NO)-mediated endothelium-dependent dilation and oxidative stress. Despite the promising evidence in pre-clinical models, there have been no reports on the efficacy of NMN supplementation in humans. There are currently five registered clinical trials examining the role of NMN supplementation on metabolic parameters including glucose and insulin metabolism, lipid levels, body composition and hormone levels.

The intervention for this open label study will be Limitless, a supplement containing NAD+ boosting ingredients, in combination with a low carbohydrate diet. This study is a pilot study to provide information on the safety and efficacy of the intervention composed of Limitless and a low-carbohydrate diet on a population of participants that are not eligible for statin therapy. This study will inform on future research to be conducted in randomized, double-blind, placebo-controlled trials designed for chronic supplementation of the investigational product together with the diet. Vascular function will be assessed by blood pressure (BP), blood flow velocity and NO metabolites as well as examine outcomes related to NAD+ metabolism, inflammation and anti-oxidant status, glucose metabolism, lipid profile, physical performance, quality of life and safety. Dietary strategies to modify hypertension have been used as part of standard of care, including the Dietary Approaches to Stop Hypertension (DASH) diet. Other dietary interventions have been used to reduce BP and improve other cardiometabolic markers in otherwise healthy adults. Indeed, both low-carbohydrate and low-fat dietary interventions have been found to reduce systolic BP (SBP) and diastolic BP (DBP) . It is acknowledged that both dietary strategies may be beneficial to this population, however we have selected a low carbohydrate diet as this is hypothesized to be more compatible with the investigational product, Limitless, as a high-carbohydrate diet negates the potential benefits of the supplement. For example, the blood-sugar mediating effects of Berberine, are countered by the blood-sugar spike caused by a carbohydrate rich diet. The carbohydrate rich diet is thought to be one contributor to high blood pressure, therefore a low carbohydrate diet in combination with the supplement is hypothesized to produce beneficial improvements in blood pressure while promoting factors that support restoration of healthy blood flow and oxygen delivery in the body.

Normal-standard-of-care is the recommendation in place for medical practitioners in the management of hypertension prior to the introduction of prescription medication plans. According to the most recent report from the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines, lifestyle modifications are recommended prior to prescribing anti-hypertensives. In Hypertension Canada's 2020 Comprehensive Guidelines for Prevention, Diagnoses, Risk Assessment, and Treatment of Hypertension in Adults and Children, patients who are low risk, defined as having no other target organ or cardiovascular risk factors suggest an initiation of anti-hypertensive therapy when systolic SBP is ≥ 160 mmHg, or diastolic DBP is ≥ 100 mmHg.

Participants in this study represent a target population who would benefit from safe and efficacious nutraceuticals for regulation of BP without the added burden of side effects that are associated with angiotensin converting enzyme (ACE) inhibitors thus limiting the complexities of polypharmacy. The current study population therefore allows for hypertensives to be enrolled if they are found to be ineligible for therapeutic plans that required prescription medication of ACE inhibitors. Participants will be assessed on a case-by-case basis to ensure that commodities and concomitant medications that may impact the safe of a passage of a participant thought this study will be monitored. Significant metabolic or physiological conditions that may affect vascular function, inflammation or glucose metabolism will be excluded. As well, an extensive list of exclusions in place will ensure that eligibility is based on establishing health and each participants' eligibility will be overseen by the Medical Director. Participants aged 45 to 65 years will be considered for enrolment to avoid complications related to advanced age and a body mass index (BMI) of and up to 32.9 kg/m2 will eliminate confounders related to advanced obesity. Sex-specific waist circumference cut-offs of less than 102 cm in men and 88 cm in women will be used to exclude individuals with an increased risk for obesity-related diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 45 and 65 years of age, inclusive
2. BMI between 20.0-32.5 + 0.1 kg/m2, inclusive
3. Waist circumference < 102 cm (40 inches) in men and < 88 cm (35 inches) in women
4. Individuals with mild hypertension (seated resting systolic blood pressures between 120-150 mmHg (inclusive) and diastolic blood pressure ≤ 95 mmHg at screening) and eligible for normal-standard-of-care, as per QI.
5. Female participant is not of child-bearing potential, defined as females who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening

   Or,

   Females of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
6. Ability to complete six-minute walk and treadmill VO2 max tests
7. Agrees to adhere to dietary guidelines and to maintain current activity level throughout the study
8. Agrees to avoid caffeine consumption 8-hours prior to in-clinic visits
9. Provided voluntary, written, informed consent to participate in the study
10. Healthy as determined by medical history, laboratory results, and EKG, as assessed by Qualified Investigator (QI)

Exclusion Criteria:

1. Women who are pregnant, breast feeding, or planning to become pregnant during the study
2. Allergy, sensitivity, or intolerance to the investigational product's active or inactive ingredients
3. Individuals who follow a vegetarian or vegan diet
4. Current use of lipid lowering medications, antihypertensive medications or prescribed medications that may affect NO synthesis as assessed by QI
5. Current use of over-the-counter medications and supplements containing the ingredients in the IP or derivatives unless willing to washout
6. Unstable metabolic disease or chronic diseases as assessed by the QI
7. Current or history of any significant diseases of the gastrointestinal tract as assessed by the QI
8. Type I or Type II diabetes
9. Significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case-by-case basis
10. History of or current diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones in participants who are symptom free for 6 months
11. Self-reported confirmation of current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
12. Major surgery in the past 3 months or individuals who have planned surgery during the course of the study. Participants with minor surgery will be considered on a case-by-case basis by the QI
13. Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
14. Individuals with an autoimmune disease or are immune-compromised
15. Self-reported confirmation of a HIV-, Hepatitis B- and/or C-positive diagnosis
16. Self-reported confirmation of blood/bleeding disorders
17. Use of medical cannabinoid products
18. Chronic use of cannabinoid products as assessed by QI on a case-by-case basis
19. Use of tobacco products within 6 months of baseline as assessed by the QI
20. Alcohol intake >2 standard drinks per day
21. Alcohol or drug abuse within the last 12 months
22. Blood donation 30 days prior to screening, during the study, or a planned donation within 30 days of the last study visit
23. Participation in other clinical research studies within 30 days of enrollment, as assessed by the QI
24. Clinically significant abnormal laboratory results at screening as assessed by the QI
25. Individuals who are unable to give informed consent
26. Any other condition, including self-reported confirmation of medical or neuropsychological condition and/or cognitive impairment, that in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures, or pose significant risk to the participant

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Changes to blood pressure from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to blood pressure will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet
Changes to forearm blood flow velocity from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to forearm blood flow will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet
Changes to plasma L-arginine from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to plasma L-arginine will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet
Changes to oral nitric oxide from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to oral nitric oxide will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet
Changes to blood nitrate from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to blood nitrate will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet
Changes to blood peroxynitrite levels from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to blood peroxynitrite levels will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet

SECONDARY OUTCOMES:
Changes to plasma nicotinamide from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to plasma nicotinamide levels will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet
Changes to blood urea from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to blood urea levels will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet
Changes to C-reactive protein from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to C-reactive protein levels will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet
Changes to homocysteine from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to homocysteine levels will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet
Changes to glutathione from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to glutathione levels will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet
Changes to triglycerides from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to triglycerides levels will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet
Changes to total cholesterol from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to total cholesterol levels will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet
Changes to high-density lipoprotein cholesterol from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to high-density lipoprotein cholesterol levels will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet
Changes to non high-density lipoprotein cholesterol from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to non high-density lipoprotein cholesterol levels will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet
Changes to low-density lipoprotein cholesterol from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to low-density lipoprotein cholesterol levels will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet
Changes to triglyceride:high-density lipoprotein cholesterol ratio from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to triglyceride:high-density lipoprotein cholesterol ratio will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet
Changes to total cholesterol:high-density lipoprotein cholesterol ratio from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to total cholesterol:high-density lipoprotein cholesterol ratio will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet
Changes to low-density lipoprotein cholesterol:high-density lipoprotein cholesterol ratio from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to low-density lipoprotein cholesterol:high-density lipoprotein cholesterol ratio will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet
Changes to blood glucose from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to blood glucose levels will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet
Changes to blood ketone levels from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to blood ketone levels will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet
Changes to blood lactic acid levels from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to blood lactic acid levels will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet
Changes to resting VO2 from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to resting VO2 levels will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet
Changes to submaximal VO2 from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to submaximal VO2 levels will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet. Changes to VO2 max will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet. Participants will be instructed to warm up on the treadmill first for five minutes at a leisurely walking pace. Participants will complete a modified Bruce Protocol on the treadmill until voluntary exhaustion by the participant. This protocol will be modified from the American College of Sports Medicine. Handrail use should be minimized during testing. Following completion of the test participants will be instructed to cool down on the treadmill for five minutes at a leisurely walking pace. Submaximal VO2 will be measured using the CardioCoach CO2 during the test and time to exhaustion will be recorded.
Changes to VO2 max from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to VO2 max will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet. Participants will be instructed to warm up on the treadmill first for five minutes at a leisurely walking pace. Participants will complete a modified Bruce Protocol on the treadmill until voluntary exhaustion by the participant. This protocol will be modified from the American College of Sports Medicine. Handrail use should be minimized during testing. Following completion of the test participants will be instructed to cool down on the treadmill for five minutes at a leisurely walking pace. Maximal VO2 will be measured using the CardioCoach CO2 during the test and time to exhaustion will be recorded.
Changes to time to exhaustion from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to time to exhaustion will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet
Changes to six-minute walk test from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to six-minute walk test will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet
Changes to quality of life from baseline to Day 30 post-supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes to quality of life will be reported from baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet. Quality of life assessed by the SF-36 Quality of Life Questionnaire. The RAND SF-36 questionnaire is a set of generic, coherent, and easily administered quality-of-life measures These measures will rely upon participant self-reporting to capture an overall indication of health-related quality of life. The SF-36 measures eight scales: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. The scores range from 0 to 100 where higher scores indicate a better state of health.
Changes to blood pressure from pre- to 2.5-hours after acute dose supplementation with Limitless in addition to a low carbohydrate diet at baseline and at Day 30 | 30 days
  Changes to blood pressure will be reported from pre- to 2.5-hours after acute dose supplementation from baseline and compared to day 30 post-supplementation with Limitless.
Changes to forearm blood flow velocity from pre- to 2.5-hours after acute dose supplementation with Limitless at baseline and at Day 30 | 30 days
  Changes to forearm blood flow velocity will be reported from pre- to 2.5-hours after acute dose supplementation from baseline and compared to day 30 post-supplementation with Limitless.
Changes to oral nitric oxide from pre- to 2.5-hours after acute dose supplementation with Limitless at baseline and at Day 30 | 30 days
  Changes to oral nitric oxide levels will be reported from pre- to 2.5-hours after acute dose supplementation from baseline and compared to day 30 post-supplementation with Limitless.
Changes to L-arginine from pre- to 2.5-hours after acute dose supplementation with Limitless at baseline and at Day 30 | 30 days
  Changes to plasma L-arginine levels will be reported from pre- to 2.5-hours after acute dose supplementation from baseline and compared to day 30 post-supplementation with Limitless.
Changes to blood nitrate from pre- to 2.5-hours after acute dose supplementation with Limitless at baseline and at Day 30 | 30 days
  Changes to blood nitrate levels will be reported from pre- to 2.5-hours after acute dose supplementation from baseline and compared to day 30 post-supplementation with Limitless.
Changes to peroxynitrite from pre- to 2.5-hours after acute dose supplementation with Limitless at baseline and at Day 30 | 30 days
  Changes to peroxynitrite levels will be reported from pre- to 2.5-hours after acute dose supplementation from baseline and compared to day 30 post-supplementation with Limitless.
Changes to plasma nicotinamide from pre- to 2.5-hours after acute dose supplementation with Limitless at baseline and at Day 30 | 30 days
  Changes to plasma nicotinamide levels will be reported from pre- to 2.5-hours after acute dose supplementation from baseline and compared to day 30 post-supplementation with Limitless.
Changes to blood urea from pre- to 2.5-hours after acute dose supplementation with Limitless at baseline and at Day 30 | 30 days
  Changes to blood urea levels will be reported from pre- to 2.5-hours after acute dose supplementation from baseline and compared to day 30 post-supplementation with Limitless.
Changes to C-reactive protein from pre- to 2.5-hours after acute dose supplementation with Limitless at baseline and at Day 30 | 30 days
  Changes to C-reactive protein levels will be reported from pre- to 2.5-hours after acute dose supplementation from baseline and compared to day 30 post-supplementation with Limitless.
Changes to homocysteine from pre- to 2.5-hours after acute dose supplementation with Limitless at baseline and at Day 30 | 30 days
  Changes to homocysteine levels will be reported from pre- to 2.5-hours after acute dose supplementation from baseline and compared to day 30 post-supplementation with Limitless.
Changes to glutathione from pre- to 2.5-hours after acute dose supplementation with Limitless at baseline and at Day 30 | 30 days
  Changes to glutathione levels will be reported from pre- to 2.5-hours after acute dose supplementation from baseline and compared to day 30 post-supplementation with Limitless.
Changes to blood pressure from pre- to post-physical performance tests (treadmill) at baseline and at day 30 post-supplementation with Limitless in addition to a low carbohydrate diet. | 30 days
  Changes to blood pressure will be reported from pre- to post-physical performance tests at baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet. Participants will be instructed to warm up on the treadmill first for five minutes at a leisurely walking pace. Participants will complete a modified Bruce Protocol on the treadmill until voluntary exhaustion by the participant. This protocol will be modified from the American College of Sports Medicine. Handrail use should be minimized during testing. Following completion of the test participants will be instructed to cool down on the treadmill for five minutes at a leisurely walking pace.
Changes to blood pressure from pre- to post-physical performance tests (six-minute walk test) at baseline and at day 30 post-supplementation with Limitless in addition to a low carbohydrate diet. | 30 days
  Changes to blood pressure will be reported from pre- to post-physical performance tests (six-minute walk test) at baseline and compared to day 30 post-supplementation with Limitless in addition to a low carbohydrate diet. A distance of 15 meters will be marked on the floor of the hallway and markers will be placed at each end of the course. The test will consist of the subject walking the length of the course, pivoting briskly at the end and returning to the starting point. The subject will complete as many laps of the course as possible over six minutes. The clinical coordinator will provide encouragement and time updates at 1-minute intervals over the length of the 6 minutes. At the 6-minute mark the subject will be asked to stop where they are standing and a clinical coordinator will calculate the distance that was walked in meters.
Product tolerability following 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Product tolerability will be assessed by the Product Tolerability Questionnaire at day 30 post supplementation with Limitless in addition to a low carbohydrate diet.
Product tolerability following 15 day supplementation with Limitless in addition to a low carbohydrate diet | 15 days
  Product tolerability will be assessed by the Product Tolerability Questionnaire at day 15 post supplementation with Limitless in addition to a low carbohydrate diet..
Product tolerability at baseline following supplementation with Limitless | baseline
  Product tolerability will be assessed by the Product Tolerability Questionnaire at at baseline post supplementation with Limitless.

OTHER OUTCOMES:
Incidence of pre-emergent adverse events following 30-day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Number of pre-emergent adverse events will be determined to calculate the incidence.
Incidence of post-emergent adverse events following 30-day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Number of post-emergent adverse events will be determined to calculate the incidence.
Changes in heart rate following 30-day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Changes in heart rate after 30-day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline.
Number of Participants With Abnormal Electrocardiogram (EKG) Readings After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  EKG reports will be analysed after 30 days supplementation with Limitless in addition to a low carbohydrate diet and compared to baseline. All EKGs will be assessed by the Qualified Investigator on a case-by-case basis to determine if they were normal or abnormal based on the full clinical picture and patient details. Number of participants with clinically relevant abnormal EKGs will be recorded.
Change in Aspartate Aminotransferase After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Change in aspartate aminotransferase after 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline.
Change in Alanine Aminotransferase After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Change in Alanine Aminotransferase After 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline.
Change in alkaline phosphatase After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Change in alkaline phosphatase After 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline.
Change in Total Bilirubin After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30
  Change in total bilirubin After 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline.
Change in creatinine After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Change in creatinine After 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline.
Change in Sodium Electrolyte Levels After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Change in Sodium Electrolyte Levels After 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline.
Change in Potassium Electrolyte Levels After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Change in Potassium Electrolyte Levels after 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline.
Change in Chloride Electrolyte Levels After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Change in Chloride Electrolyte Levels after 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline.
Change in Estimated Glomerular Filtration Rate (eGFR) After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Change in eGFR after 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline.
Change in White Blood Cell (WBC) Count After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Change in WBC count after 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline
Change in Amount of Neutrophils After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Change in amount of neutrophils after 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline
Change in Amount of Lymphocytes After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Change in amount of lymphocytes after 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline
Change in Amount of Monocytes After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Change in amount of monocytes after 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline
Change in Amount of Eosinophils After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Change in amount of eosinophils after 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline
Change in Amount of Basophils After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Change in amount of basophils after 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline
Change in Amount of immature granulocytes After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Change in amount of immature granulocytes after 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline
Change in Amount of nucleated RBC After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Change in amount of nucleated RBC after 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline
Change in Red Blood Cell (RBC) Count After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Change in RBC count after 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline
Change in Hemoglobin Levels After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Change in Hemoglobin Levels after 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline.
Change in Hematocrit Levels After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Change in Hematocrit Levels after 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline.
Change in Platelet Count After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Change in platelet count after 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline.
Change in Mean Corpuscular Volume (MCV) After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Change in MCV after 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline.
Change in Mean Corpuscular Hemoglobin (MCH) After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Change in MCH after 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline.
Change in Mean Corpuscular Hemoglobin concentration (MCHC) After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Change in MCHC after 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline.
Change in Red Cell Distribution Width (RDW) After 30 day supplementation with Limitless in addition to a low carbohydrate diet | 30 days
  Change in RDW after 30 day supplementation with Limitless in addition to a low carbohydrate diet compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada